CLINICAL TRIAL: NCT07358754
Title: The Relationship Between Serum S100B and Brain-Derived Neurotrophic Factor (BDNF) Levels and Central Sensitization and Sleep Quality in Patients With Fibromyalgia
Brief Title: The Relationship Between Serum S100B and Brain-Derived Neurotrophic Factor
Acronym: S100B-BDNF
Status: Not yet recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Karakuzu Güngör, Physical Medicine and Rehabilitation Specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KSS-EAH-FMS-S100B-BDNF-2026
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected from all participants at a single time point. Serum will be separated and used for the measurement of S100B and brain-derived neurotrophic factor (BDNF) levels. No genetic or DNA analyses will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fibromyalgia Group: Female patients aged 18-50 years diagnosed with fibromyalgia according to the 2016 American College of Rheumatology criteria.
  Interventions: Other: No Intervention (Observational Study)
- Healthy Control Group: Age- and sex-matched healthy female volunteers without fibromyalgia or chronic widespread pain.
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — This is an observational study with no therapeutic or diagnostic intervention. Participants will undergo a single-time-point clinical assessment and venous blood sampling for biomarker measurement only.

SUMMARY:
Fibromyalgia is a chronic pain syndrome characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and cognitive symptoms. Central sensitization is considered a key mechanism in the pathophysiology of fibromyalgia; however, the underlying biological markers have not been fully clarified.

Brain-derived neurotrophic factor (BDNF) and S100B protein have been suggested to play roles in neuroinflammation and central pain processing. This observational, cross-sectional study aims to evaluate serum S100B and BDNF levels in patients with fibromyalgia and to investigate their relationship with central sensitization and sleep quality. Serum biomarker levels and clinical assessment scales will be compared between patients with fibromyalgia and healthy controls.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain syndrome characterized by widespread musculoskeletal pain, fatigue, sleep disturbances, and cognitive complaints. Central sensitization, defined as increased responsiveness of the central nervous system to sensory stimuli, is considered a core mechanism in the pathophysiology of fibromyalgia. However, the biological processes underlying central sensitization and associated clinical features such as sleep disturbances remain incompletely understood.

Brain-derived neurotrophic factor (BDNF) is a neurotrophin involved in synaptic plasticity, neuronal survival, and pain modulation, and has been suggested to be associated with central sensitization. S100B is a calcium-binding protein predominantly released by astrocytes and is considered a peripheral marker of neuroinflammation and glial activation. Alterations in serum levels of BDNF and S100B have been reported in chronic pain conditions, including fibromyalgia.

This observational, cross-sectional study aims to evaluate serum S100B and BDNF levels in patients diagnosed with fibromyalgia according to the 2016 American College of Rheumatology criteria and to investigate their relationship with central sensitization and sleep quality. A healthy control group matched for age and sex will be included for comparative analysis.

All participants will undergo a single-time-point assessment, including collection of demographic and clinical data. Blood samples will be obtained to measure serum S100B and BDNF levels using standard laboratory methods. Central sensitization will be assessed using the Central Sensitization Inventory, while sleep quality will be evaluated using the Pittsburgh Sleep Quality Index. Additional clinical assessments will include the Fibromyalgia Impact Questionnaire, Beck Depression Inventory, and Beck Anxiety Inventory.

The study does not involve any therapeutic intervention or randomization. The findings are expected to contribute to a better understanding of the biological correlates of central sensitization and sleep disturbances in fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 50 years

Diagnosis of fibromyalgia according to 2016 American College of Rheumatology (ACR) criteria

Symptoms present for at least 3 months

Ability to understand and complete study questionnaires

Provision of written informed consent

For healthy controls:

No diagnosis of fibromyalgia or chronic widespread pain

No known systemic disease

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is NOT based on self-representation of gender identity.
Study Population: Presence of any systemic disease (hematologic, endocrine, rheumatologic, renal, cardiovascular, gastrointestinal, or respiratory) Active infection History of malignancy Major surgery or trauma within the last 1 year Any treatment for fibromyalgia within the last 3 months Pregnancy or breastfeeding Smoking Vitamin D deficiency
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Association between serum S100B and serum BDNF | Baseline
  Serum S100B and serum BDNF concentrations will be measured from venous blood samples and the strength of association between the two biomarkers will be analyzed

SECONDARY OUTCOMES:
Correlation of serum S100B and BDNF with Central Sensitization Inventory (CSI) | Baseline
  Serum S100B and BDNF levels will be correlated with CSI total score to evaluate biomarker association with central sensitization severity.
Correlation of serum S100B and BDNF with Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Serum S100B and BDNF levels will be correlated with PSQI total score to evaluate association with sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karakuzu Güngör, M.D, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly. De-identified aggregate data may be made available upon reasonable request from the corresponding author after publication of the study results.